CLINICAL TRIAL: NCT02432742
Title: A Randomised, Multi-center, Evaluator-blinded Study in China to Evaluate the Efficacy and Safety of Restylane Perlane Compared to Restylane for Correction of Moderate to Severe Nasolabial Folds
Brief Title: Efficacy and Safety of Restylane Perlane Compared to Restylane for Correction of Moderate and Severe Nasolabial Folds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 43CH1408
Record Dates: First submitted 2015-04-23; First posted 2015-05-04 (Estimated); Results first posted 2020-12-23 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2021-02

CONDITIONS: Nasolabial Folds in Chinese Population
Keywords: hyaluronic acid, comparative study, NLF

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Restylane Perlane (Experimental): Single injection and optional touch up injection with Restylane Perlane in NLF
  Interventions: Device: Restylane Perlane
- Restylane (Active Comparator): Single injection and optional touch up injection with Restylane in NLF
  Interventions: Device: Restylane

INTERVENTIONS:
Device: Restylane Perlane — Intradermal injection
  Arms: Restylane Perlane
Device: Restylane — Intradermal injection
  Arms: Restylane

SUMMARY:
The purpose of this study is to determine the safety and efficacy of using Restylane Perlane compared to Restylane for correction of moderate to severe nasolabial folds (NLF) in a Chinese population.

ELIGIBILITY:
Inclusion Criteria:

* Chinese origin
* Subjects intent to undergo correction of both NLFs with a Wrinkle Severity Rating Scale (WSRS) of 3 on both side or 4 on both side.
* Subjects willing to abstain from other facial plastic surgical or cosmetic procedures during the study period.
* Singed Informed Consent

Exclusion Criteria:

* Subjects with traumatic scars or ongoing active skin disease in the area to be treated
* Permanent inplant or filler, including fat injection placed in the area to be treated
* Previous tissue augmentation therapy in the NLFs with non-permanent filler within 12 months prior to inclusion
* Any medical condition in the opinion of the treating investigator who will make the subject unsuitable for inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-05; Primary Completion 2016-03 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Q-Med AB, Study Director — Galderma R&D
Locations (3):
- China (3):
  - Beijing
  - Wuhan
  - Zhejiang

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Restylane Perlane in One NLF and Restylane in the Other NLF: Single injection and optional touch up injection with Restylane Perlane in one nasolabial fold (NLF) and single injection and optional touch up injection with Restylane in the other NLF (split-face design).
  Restylane Perlane: Intradermal injection Restylane: Intradermal injection
Period: Overall Study
Arm/Group | Restylane Perlane in One NLF and Restylane in the Other NLF
Started | 100
Completed | 95
Not Completed | 5

BASELINE CHARACTERISTICS:
Groups:
- Restylane Perlane in One NLF and Restylane in the Other NLF: Single injection and optional touch up injection with Restylane Perlane in one NLF and single injection and optional touch up injection with Restylane in the other NLF (split-face design).
  Restylane Perlane: Intradermal injection, Restylane: Intradermal injection
Arm/Group | Restylane Perlane in One NLF and Restylane in the Other NLF
Number analyzed (Participants) | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 100
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Sex: Female | 98
  Sex: Male | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Han Chinese | 97
  Ethnicity: Other (Manchu, Tujia, Hui) | 3
Region of Enrollment [Count of Participants; unit: Participants]
  China | 100
WSRS score of either 3 on both sides or 4 on both sides as assessed by an Independent Evaluator [Count of Participants; unit: Participants] — The Wrinkle Severity Rating Scale (WSRS) is a 5-graded scale with grades 1-5 ranging from absent (1) to extreme (5). A clinical significant improvement is defined as at least 1 grade improvement (lowering in grade).
  Participants | 100

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Wrinkle Severity Rating Scale (WSRS) at 6 Months
Description: The Wrinkle Severity Rating Scale (WSRS) is a 5-graded scale with grades 1-5 ranging from absent (1) to extreme (5). A clinical significant improvement is defined as at least 1 grade improvement (lowering in grade).
Time Frame: 6 months
Population: Split-face design; 100 participants received treatment with Restylane Perlane in one NLF and treatment with Restylane in the other NLF.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Restylane Perlane NLFs: Single injection and optional touch up injection with Restylane Perlane in NLF
  Restylane Perlane: Intradermal injection
- Restylane NLFs: Single injection and optional touch up injection with Restylane in NLF
  Restylane: Intradermal injection
Arm/Group | Restylane Perlane NLFs | Restylane NLFs
Number analyzed (Participants) | 100 | 100
units on a scale | -0.03 (0.03) | 0.03 (0.03)

ADVERSE EVENTS:
Arm/Group | Restylane Perlane in One NLF and Restylane in the Other NLF
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 2/100
Other Adverse Events (participants affected / at risk) | 16/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Restylane Perlane in One NLF and Restylane in the Other NLF (N=100)
Multi organ failure, infection (Infections and infestations) | 1 (1) — Not related to study product or study product injection procedure
Bladder lesion excision (Surgical and medical procedures) | 1 (1) — Not related to study product or study product injection procedure
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Restylane Perlane in One NLF and Restylane in the Other NLF (N=100)
Nasopharyngitis (Infections and infestations) | 9 (10) — Not related to study product or study product injection procedure: Frequency Threshold > 5%
Upper respiratory tract infection (Infections and infestations) | 5 (5) — Not related to study product or study product injection procedure: Frequency Threshold > 5%
Implant site bruising (General disorders) | 1 (1) — Restylane Perlane: Intensity of related adverse event
Implant site bruising (General disorders) | 1 (1) — Restylane: Intensity of related adverse event

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes